CLINICAL TRIAL: NCT03171142
Title: Effect of Heliox on Infants With Respiratory Syncytial Virus Acute Bronchiolitis-A Revisit Study
Brief Title: Effect of Heliox on RSV Bronchiolitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wael Seliem (Other)
Responsible Party: Sponsor-Investigator, Wael Seliem, Associated Professor, Mansoura University Children Hospital
Organization: Mansoura University Children Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R/17.01.55
Record Dates: First submitted 2017-05-24; First posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: RSV Infection; Acute Bronchiolitis
Keywords: Heliox
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — heliox; Air

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heliox group (Active Comparator): receive Helium oxygen mixture 21:79 via nasal cannula 2L/min
  Interventions: Drug: Heliox
- Air group (Active Comparator): receive oxygen 21%via nasal cannula 2L/min
  Interventions: Drug: Air

INTERVENTIONS:
Drug: Heliox — Heliox (21:79) via nasal cannula 2 litter per minutes
  Arms: Heliox group
Drug: Air — Air 21% via nasal cannula 2 litter per minutes
  Arms: Air group

SUMMARY:
Helium is an inert gas with a density almost one-seventh of that of air. Based on its properties breathing a mixture of helium and oxygen (heliox) will lead to a reduction in resistance through narrowed airways and consequently decreases the work of breathing. Participating infants with RSV acute bronchiolitis will be supplied with heliox (ration of 21 oxygen and 79 helium) delivered through a flow nasal cannula to evaluate heliox effect in improving their oxygenation. Heliox will act as an additive therapy to improve oxygenation in patients with lower respiratory tract infection caused by respiratory Syncytial Virus (RSV) and will decrease the need for more complicated therapies.

ELIGIBILITY:
Inclusion Criteria:

* Age fro 1 month till 2 years
* RSV acute bronchiolitis without any supplemental oxygen.

Exclusion Criteria:

* oxygen supplement or mechanical ventilation requirement
* congenital anomalies of the heart
* chronic lung disease including bronchopulmonary dysplasia
* Failure to obtain an informed consent.

Ages: 1 Month to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2016-08-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Improvement in oxygenation | change from baseline at 24 hours after treatment
  Arterial blood samples will be withdrawn through an arterial stab to determine partial pressure of arterial oxygen (PaO2)

SECONDARY OUTCOMES:
improvement of respiratory distress | change from baseline at 24 hours after treatment
  measured by the Modified Wood's Clinical Asthma Score